CLINICAL TRIAL: NCT01546545
Title: Testing Whether Insulin Resistance Varies Throughout a Day A Pilot Study
Brief Title: Insulin Variance Throughout the Day
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Jenny Craig, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PBRC 11021
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-08

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — IV Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin Sensitivity in Pre-Diabetic Population: Healthy participants between the age of 18 and 70 years with fasting blood sugar that is between normal and diabetes.

SUMMARY:
This study is designed to determine whether the sensitivity of a participant's insulin varies from the morning to the evening.

DETAILED DESCRIPTION:
Study visit 1: about 16 hours - The participant will arrive to the visit fasting.

The participant will have an oral glucose tolerance test which takes about 3 ½ hours.

An IV line will be placed in the participant's arm vein for blood draw purposes and will remain there throughout the testing. A blood sample will be drawn 15 minutes and just before the participant will drink a sugar solution consisting of 75 grams of glucose. Blood will be drawn at specific times after the participant consumes the drink.

The participant will have a second oral glucose tolerance test which takes about 3 ½ hours. An IV line will be placed in the participant's arm vein for blood draw purposes and will remain there throughout the testing. A blood sample will be drawn 15 minutes and just before the participant drinks a sugar solution. Blood will be drawn at specific times after the participant consumes the drink.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy male or female
* Have a fasting blood sugar that is between normal and diabetes.
* Are between 18 and 70 years of age, inclusive.

Exclusion Criteria:

* Are pregnant or breast-feeding a child
* Take a medication for diabetes
* Take a medication like cortisone that can change your blood sugar.
* Take a medication chronically that has not been at a stable dose for at least 1 month
* Take medication for psychosis that is known to change timing in the day - night cycle

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants with blood sugar between normal and diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gimble, MD, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Sensitivity in Pre-Diabetic Population
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Circadian Variablity of insulin sensitivity in a pre-diabetic population.
Arm/Group | Insulin Sensitivity in Pre-Diabetic Population
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Glucose Tolerance Between Morning at 7:00 AM and Evening at 7:00 PM
Description: This study designed to determine whether glucose tolerance varies from the morning to the evening. The test is useful in the diagnosis of diabetes and pre diabetes. Oral Glucose Tolerance Testing (OGTT) provides details about how quickly glucose is absorbed into the bloodstream for use by body cells as energy. The rate of glucose clearance depends on the amount of glucose consumed and insulin levels. Once the participant drink a glucose-rich beverage, blood will be drawn at two and three hour points, and tested to see how effective the body metabolizes blood glucose.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Morning OGTT at 7:00 AM; Evening OGTT at 7:00 PM: Ten subjects with prediabetes completed oral glucose tolerance tests at 7:00 AM and 7:00 PM on the same day. Lipids and hormones were also measured.
Arm/Group | Morning OGTT at 7:00 AM | Evening OGTT at 7:00 PM
Number analyzed (Participants) | 10 | 10
mg/dl | 163 (62) | 203 (71)
Statistical Analysis 1: Comparison: Morning OGTT at 7:00 AM vs Evening OGTT at 7:00 PM; Test type: Non-Inferiority or Equivalence — No power calculation was performed. This was the first pilot and feasibility study. This data will be used to power future studies; p = 0.02, t-test, 2 sided

2. Primary Outcome: Difference Between Morning at 7:00 AM and Evening at 7:00 PM 2-hour AUC Insulin Levels During an OGTT
Description: This study designed to determine whether insulin levels vary from the morning at 7:00 AM to the evening at 7:00 PM. The test is useful in the diagnosis of diabetes and pre diabetes. Oral Glucose Tolerance Testing (OGTT) provides details about how quickly glucose is absorbed into the bloodstream for use by body cells as energy. The rate of glucose clearance depends on the amount of glucose consumed and the amount of insulin in the body. Once the participant drink a glucose-rich beverage, blood will be drawn at two and three hour points, and tested to see how effective the body metabolizes blood glucose.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: UI*hr/L
Groups:
- AUC Insulin Levels During an OGTT at 7:00 AM; AUC Insulin Levels During an OGTT at 7:00 PM: Ten subjects with prediabetes completed oral glucose tolerance tests at 7:00 AM and 7:00 PM on the same day. Lipids and hormones were also measured.
Arm/Group | AUC Insulin Levels During an OGTT at 7:00 AM | AUC Insulin Levels During an OGTT at 7:00 PM
Number analyzed (Participants) | 10 | 10
UI*hr/L | 69.8 (40.2) | 87.4 (37.6)
Statistical Analysis 1: Comparison: AUC Insulin Levels During an OGTT at 7:00 AM vs AUC Insulin Levels During an OGTT at 7:00 PM; Test type: Non-Inferiority or Equivalence — No power calculation was performed. This was a pilot and feasibility study; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Insulin Sensitivity in Pre-Diabetic Population
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Sensitivity in Pre-Diabetic Population (N=11)
Nausea and vomitting during OGTT (Gastrointestinal disorders) | 1 — One participant got nauseous and vomitted during the Oral Glucose Tolerance Testing. This is an infrequent known side effect of the test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes